CLINICAL TRIAL: NCT01972581
Title: Neurocognitive Visual Reaction Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: High Point University (Other)
Responsible Party: Principal Investigator, Kevin Ray Ford, Director, Biomechanics Laboratory, High Point University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: HBAPL-201309-191
Record Dates: First submitted 2013-10-21; First posted 2013-10-30 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Reaction Time
Keywords: neurocognitive visual reaction training; baseball

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reaction Time Training (Experimental)
  Interventions: Other: Reaction Time Training
- Control (No Intervention)

INTERVENTIONS:
Other: Reaction Time Training
  Arms: Reaction Time Training

SUMMARY:
Incorporating neurocognitive visual reaction training has been shown to increase bating performance in collegiate baseball players. However, poor methodology, such as lack of a control group and use of an unreliable outcome measure, limit the strength of the previous study. Therefore the purpose of this study is to determine the effects of neurocognitive visual reaction training on reaction time and coordination in an athletic population.

The purpose of this study is to determine the effects of neurocognitive visual reaction training on reaction time and coordination.

ELIGIBILITY:
Inclusion Criteria:

* subjects that participate in a structured sport team
* between the ages of 18-65
* with or without a history of mild traumatic brain injury.

Exclusion Criteria:

* subjects currently under medical supervision and not fully cleared to participate in structured sport team.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Number of colored balls correctly identified | 5 weeks

SECONDARY OUTCOMES:
Number of ball catches on alternate ball toss | 5 weeks
Reaction time on dynavision reaction board | 5 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Ford, PhD, Principal Investigator — High Point University
Locations (1):
- Human Biomechanics and Physiology Laboratory, High Point, North Carolina, United States